CLINICAL TRIAL: NCT06867354
Title: Prevalence, Determinants and Consequences of Dyspnea During Weaning in Critically Ill Obese Patients
Acronym: WEAN OBESE
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP241581; IDRCB-2024-A02501-46 (Other: ANSM)
Record Dates: First submitted 2025-01-22; First posted 2025-03-10 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Obesity; Obesity With Complications; Weaning From Mechanical Ventilation in Care Unit; Dyspnea
Keywords: Intensive Care Unit; Dyspnea; Mechanical Ventilation; Ventilatory Weaning; Obesity; Spontaneous Ventilation Test; Mortality
MeSH Terms: conditions — Obesity; Dyspnea

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients with (BMI of ≥30 kg/m²) obesity
- Patients without obesity

SUMMARY:
ICU patients encounter numerous discomforts, with dyspnea (the sensation of breathlessness) being among the most distressing and impactful. Unlike pain, dyspnea in ICU settings has historically received limited attention, despite its severe psychological impact. ICU clinicians often use assessment tools like the simple numerical dyspnea scale (Dyspnea-VAS) and the Respiratory Distress Observation Scale (MV-RDOS) to measure dyspnea. These scales are also utilized during the weaning process, an essential phase when patients attempt to breathe independently without ventilator assistance. Weaning is crucial for ICU patients, as delayed or unsuccessful extubation increases the risk of complications and mortality.

Obese ICU patients, often admitted due to respiratory failure, present unique challenges due to physiological changes in the respiratory system, such as reduced functional residual capacity and decreased lung compliance. These factors contribute to an increased likelihood of dyspnea and weaning complications. Approximately 50% of obese ICU patients require mechanical ventilation, and once ventilated, obese patients exhibit an elevated risk for dyspnea and ventilator weaning failure.

Understanding the prevalence, causes, and consequences of dyspnea and failure in weaning process in obese ICU patients is critical. In this study, the aim is to compare obese patients with non-obese patients in terms of dyspnea prevalence, causes and consequences as weaning failure prevalence, causes and consequences.

DETAILED DESCRIPTION:
Research Justification:

ICU patients face numerous sources of discomfort, among which dyspnea- the subjective sensation of breathlessness-stands out as especially distressing. Unlike pain, dyspnea has historically received limited attention, despite its severe psychological impact, including feelings of panic and death anxiety. Dyspnea integrates both physical and psychological suffering, often leading patients to report it as one of the most unbearable experiences, highlighting its significance for ICU caregivers. The subjective nature of dyspnea presents a diagnostic challenge, as it may occur without visible respiratory distress, which complicates detection and management. Dyspnea arises from complex mechanisms, including increased respiratory muscle load from airway resistance or thoracic compliance reduction. Additionally, dyspnea can be induced by an increased need for air due to elevated carbon dioxide levels or reduced oxygen levels, triggering chemoreceptor responses.

For ICU patients mechanically ventilated, the prevalence of dyspnea has been reported between 34 and 47%. Dyspnea assessment tools, such as the Dyspnea-VAS (Visual Analog Scale) and the MV-RDOS (Respiratory Distress Observation Scale), are employed to measure dyspnea, even in intubated patients. These tools are especially useful during ventilator weaning, a critical phase when patients transition to spontaneous breathing. The weaning process, and particularly the spontaneous breathing test (SBT), a test during which the patient breath with the assistance of the ventilator, is critical. The failure of a SBT can increase mortality risk, length of mechanical ventilation and ICU stay.

In this study, the investigators focus in obesity. The growing prevalence of obesity adds an additional layer of complexity to ICU care, as obese patients present distinct challenges during ventilation and weaning. With physiological changes such as reduced lung compliance and increased airway resistance, obese patients have an elevated risk for dyspnea and ventilator weaning complications. Obesity prevalence surged during the COVID-19 pandemic until 40% of ICU patients, and today, up to 50% of obese ICU patients require mechanical ventilation.

In ICU obese patients and mechanically ventilated, there is no assessment of dyspnea, its determinants and its impact during ventilatory weaning. The pathophysiology of dyspnea and SBT failure is complex and primarily involves cardiac function and respiratory muscle function. Pulmonary edema is found in more than half of cases and is linked to the transition from a positive pressure ventilation regime to a negative pressure regime, which creates unfavorable loading conditions for the heart. The second cause described is diaphragmatic dysfunction characterized by atrophy of the respiratory muscles which can occur rapidly under mechanical ventilation. More recently, dyspnea has been described as a cause of SBT and extubation failure in its own right. Other causes have also been described such as intensive care neuropathy, iatrogenic causes (agitation, pain), anxiety, or even impaired ventilatory control.

In addition, the consequences of dyspnea and failure of SBT as well as their management are not described, such as the duration of mechanical ventilation, mortality, length of stay, intercurrent events such as new sepsis. or the administration of new treatments during the period from weaning to extubation.

Finally, the evolution of dyspnea after successful SBT and after extubation has never been described.

The prevalence, determinants and consequences of dyspnea and failure of the first SBT as well as their management in ICU patients with obesity have never been described. Likewise, improving the diagnostic performance of the clinical criteria for SBT failure with the contribution of dyspnea scales is a real challenge in these patients.

Research Design and Methodology:

Study Type: This is a descriptive, monocentric and comparative study.

ELIGIBILITY:
Inclusion Criteria:

* Patients placed on mechanical ventilation for at least 48 hours
* On spontaneous ventilation mode with inspiratory support (only possible ventilation mode during ventilation weaning) allowing a tidal volume > 6 mL/kg and a positive end-expiratory pressure set by the attending physician between 5 and 8 cmH2O
* Decision by the attending physician to perform a spontaneous breathing trial (SBT) after verifying the prerequisites for weaning: resolution of the acute phase of the illness for which the patient is placed on invasive mechanical ventilation, low bronchial congestion, adequate cough, adequate oxygenation defined by SpO2 > 90% with FiO2 ≤ 40% and PEEP ≤ 8 cmH2O, respiratory rate ≤ 40 breaths/min, Ramsay sedation score < 4, and stable cardiovascular state (heart rate ≤ 120 beats/min, systolic blood pressure ≤ 180 mmHg, and no or minimal vasopressors [norepinephrine < 5 μg/kg/min])
* After information,no opposition from the patient or the relative (if the patient is unable to express his non opposition) to participating in the research
* Person affiliated with a social security regime or eligible
* Patient with a BMI > 30 kg/m² for those included in the case group (obesity)

Exclusion Criteria:

* Under 18 years old
* Pregnant or breastfeeding women
* Patients for whom weaning is impossible (pre-existing neuromuscular disorders, cervical spinal cord lesions)
* Patients for whom repeated dyspnea assessment is likely to be difficult (known history of cognitive or psychiatric disorders, delirium, Richmond Agitation-Sedation Scale score less than -2 or greater than 2)
* Patients under legal protection measures (guardianship, curatorship)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in intensive care under mechanical ventilation for at least 48 hours, with or without obesity (BMI > 30 kg/m²).
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-03-21 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Presence or onset of dyspnea | Baseline
  Presence or onset of dyspnea detected by the simple numerical dyspnea scale (Dyspnea-Visual Analog Scale VAS) from 0 to 10 cm , 0 means "no respiratory discomfort, no sensation of shortness of breath, no difficulty breathing" and 10 means "the worst imaginable respiratory discomfort, feeling of shortness of breath, inability to breathe" ≥ 4 before, and then at 2 minutes, 15 minutes, 30 minutes, and at the end of SBT.
  In order to describe the prevalence of dyspnea during the first SBT in obese patients hospitalized in the ICU compared to non-obese patients.

SECONDARY OUTCOMES:
Measure of the affective component of dyspnea using the simple numerical dyspnea scale | Baseline
  Measure of the affective component of dyspnea using the simple numerical dyspnea scale (Dyspnea-Visual Analog Scale VAS) from 0 to 10, 0 means "no anxiety related to dyspnea" and10 means "maximum anxiety related to dyspnea" before, and then at 2 minutes, 15 minutes, 30 minutes, and at the end of SBT, anxiety if Dyspnea-VAS > 4, in order to describe the prevalence of dyspnea during the first SBT in obese patients hospitalized in the ICU compared to non-obese patients.
: Presence or onset of dyspnea detected by the Mechanical Ventilation - Respiratory Distress Observation Scale | Baseline
  Presence or onset of dyspnea detected by the Mechanical Ventilation - Respiratory Distress Observation Scale (MV-RDOS) in mechanically ventilated in non-communicating patients from 0 to 5, 0 means no dyspnea and 5 means major dyspnea, before SBT then at 2 minutes, 15 minutes, 30 minutes, and at the end of SBT, dyspnea if MV-RDOS> 2.6, in order to describe the prevalence of dyspnea during the first SBT in obese patients hospitalized in the ICU compared to non-obese patients.
Measure of Rapid Shallow Breathing Index (RSBI) (the ratio of respiratory frequency (f) to tidal volume (TV)) measured at 1 minute of SBT > 105 breaths/min/L. | Baseline
  Measure of Rapid Shallow Breathing Index (RSBI) in order to describe the prevalence of dyspnea during the first SBT in obese patients hospitalized in the ICU compared to non-obese patients.
Measure of Pain with Visual Analog Scale (VAS) for pain from 1 to 100 mm (1 means no pain, 100 means major pain) | Baseline
  Measure of pain in order to describe the main determinants of dyspnea during the first SBT in ICU patients and affected (case) or not (control) by obesity
Research of anxiety with Hospital Anxiety and Depression Scale (HADS) from 0 to 21, 0 means no anxiety, 21 means major anxiety, anxiety if HADS > 8 | Baseline
  Research of anxiety in order to describe the main determinants of dyspnea during the first SBT in ICU patients and affected (case) or not (control) by obesity
Number of patients with Respiratory Control Impairment: | Baseline
  Number of patients with Respiratory Control Impairment in order to describe the main determinants of dyspnea during the first SBT in ICU patients and affected (case) or not (control) by obesity
Measure of the number of treatments added during SBT | Baseline
  Measure of the number of treatments added during SBT in order to describe the main determinants of dyspnea during the first SBT in ICU patients and affected (case) or not (control) by obesity
Measure of the number of patients with early cessation of SBT at the patient's request for reasons unrelated to the validated clinical objective criteria for SBT failure; | Length of the ICU hospitalization (2 months maximum)
  Measure of the number of patients with early cessation of SBT at the patient's request in order to describe the clinical and therapeutic consequences of dyspnea between the first SBT and extubation in ICU patients and affected (case) or not (control) by obesity.
Measure of number of SBT performed until extubation | Length of the ICU hospitalization (2 months maximum)
  Measure of number of SBT performed until extubation in order to describe the clinical and therapeutic consequences of dyspnea between the first SBT and extubation in ICU patients and affected (case) or not (control) by obesity.
Measure of the duration between the first SBT and the extubation | Length of the ICU hospitalization (2 months maximum)
  Measure of the duration between the first SBT and the extubation in order to describe the clinical and therapeutic consequences of dyspnea between the first SBT and extubation in ICU patients and affected (case) or not (control) by obesity.
Measure of the number of extubation failure defined by reintubation or death | Within 7 days following extubation;
  Measure of the number of extubation failure in order to describe the clinical and therapeutic consequences of dyspnea between the first SBT and extubation in ICU patients and affected (case) or not (control) by obesity.
Measure of the duration of invasive and non-invasive mechanical ventilation | Length of the ICU hospitalization (2 months maximum)
  Measure of the duration of invasive and non-invasive mechanical ventilation in order to describe the clinical and therapeutic consequences of dyspnea between the first SBT and extubation in ICU patients and affected (case) or not (control) by obesity.
Measure of the length of stay in the ICU | Length of the ICU hospitalization (2 months maximum)
  Measure of the length of stay in the ICU in order to describe the clinical and therapeutic consequences of dyspnea between the first SBT and extubation in ICU patients and affected (case) or not (control) by obesity.
Measure of number of deaths in ICU | Length of the ICU hospitalization (2 months maximum)
  Measure of number of deaths in ICU in order to describe the clinical and therapeutic consequences of dyspnea between the first SBT and extubation in ICU patients and affected (case) or not (control) by obesity.
Measure of number of intercurrent events between the clinical outcome of the first SBT and extubation | Length of the ICU hospitalization (2 months maximum)
  Measure of number of intercurrent events between the clinical outcome of the first SBT and extubation in order to describe the clinical and therapeutic consequences of dyspnea between the first SBT and extubation in ICU patients and affected (case) or not (control) by obesity.
Research of the number of treatments administered between the first SBT and extubation | Length of the ICU hospitalization (2 months maximum)
  Research of the number of treatments administered between the first SBT and extubation in order to describe the clinical and therapeutic consequences of dyspnea between the first SBT and extubation in ICU patients and affected (case) or not (control) by obesity.
Description of the prevalence of first SBT failure in ICU patients and affected (case) or not (control) by obesity. | Baseline
  SBT failure defined by the appearance of at least one of the following objective criteria
  1. Respiratory rate ≥ 35 breaths/min or an increase ≥ 50% compared to the baseline value,
  2. SpO2 ≤ 90% or PaO2 ≤ 50 mmHg with FiO2 ≥ 50%,
  3. PaCO2 > 50 mmHg,
  4. Heart rate ≥ 140 beats per minute,
  5. New supraventricular or ventricular arrhythmia,
  6. Systolic blood pressure >180 or < 90 mmHg,
  7. Altered consciousness,
  8. Signs of respiratory distress.
Measure of the number of patient with pulmonary edema during weaning | Baseline
  Measure of the number of patient with pulmonary edema during weaning in order to describe the main causes of first SBT failure.
Measure of the number of patient with acute myocardial ischemia (coronary syndrome with or without ST-segment elevation) | Baseline
  Measure of the number of patient with acute myocardial ischemia (coronary syndrome with or without ST-segment elevation):in order to describe the main causes of first SBT failure.
Measure of the number of patient with respiratory muscle impairment and diaphragmatic dysfunction | Baseline
  Measure of the number of patient with respiratory muscle impairment and diaphragmatic dysfunction in order to describe the main causes of first SBT failure.
Measure of the number of patient with critical illness neuromyopathy | Baseline
  Measure of the number of patient with critical illness neuromyopathy in order to describe the main causes of first SBT failure.
Measure of the number of patient with dyspnea | Baseline
  Measure of the number of patient with dyspnea in order to describe the main causes of first SBT failure.
Measure of the number of patient with anxiety with Hospital Anxiety and Depression Scale (HADS) from 0 to 21, 0 means no anxiety, 21 means major anxiety, anxiety if HADS > 8 | Baseline
  Measure of the number of Measure of the number of patient with anxiety in order to describe the main causes of first SBT failure.
Measure of the number of patient with respiratory control impairment: | Baseline
  Measure of the number of patient with respiratory control impairment in order to describe the main causes of first SBT failure.
Measure of the number of patient with an early cessation of the SBT at the patient's request, outside of the validated clinical objective criteria for SBT | Length of the ICU hospitalization (2 months maximum)
  Measure of the number of patient with an early cessation of the SBT at the patient's request, outside of the validated clinical objective criteria for SBT failure in order to describe the clinical and therapeutic consequences of the failure of the first SBT until extubation
Measure of Number of SBT performed until extubation | Length of the ICU hospitalization (2 months maximum)
  Measure of the number of Number of SBT performed until extubation in order to describe the clinical and therapeutic consequences of the failure of the first SBT until extubation
Measure of the Delay between the date of the first SBT and the date of extubation | Length of the ICU hospitalization (2 months maximum)
  Measure of the delay between the date of the first SBT and the date of extubation in order to describe the clinical and therapeutic consequences of the failure of the first SBT until extubation
Measure of the number of patient with an extubation failure defined by reintubation or death | Length of the ICU hospitalization (2 months maximum)
  Measure of the number of patient with an extubation failure defined by reintubation or death within 7 days following extubation in order to describe the clinical and therapeutic consequences of the failure of the first SBT until extubation
Measure of the duration of invasive and non-invasive mechanical ventilation | Length of the ICU hospitalization (2 months maximum)
  Measure of the duration of invasive and non-invasive mechanical ventilation in order to describe the clinical and therapeutic consequences of the failure of the first SBT until extubation
Measure of Duration of stay in the ICU | Length of the ICU hospitalization (2 months maximum)
  Measure of Duration of stay in the ICU in order to describe the clinical and therapeutic consequences of the failure of the first SBT until extubation
Measure of the number of deaths in the ICU | Length of the ICU hospitalization (2 months maximum)
  Measure of the number of deaths in the ICU in order to describe the clinical and therapeutic consequences of the failure of the first SBT until extubation
Measure of the number of Intercurrent events between the clinical outcome of the first SBT and extubation | Length of the ICU hospitalization (2 months maximum)
  Measure of the number of Intercurrent events between the clinical outcome of the first SBT and extubation in order to describe the clinical and therapeutic consequences of the failure of the first SBT until extubation
Evaluate the contribution of combining the dyspnea scales measured during SBT with the usual clinical criteria to predict the diagnosis of SBT failure. | Length of the ICU hospitalization (2 months maximum)
  Contribution of combining the dyspnea scales measured during SBT with the usual clinical criteria to predict the diagnosis of SBT failure (area under the curve, sensitivity, specificity, likelihood ratio).
Description of the evolution of dyspnea after extubation. | Length of the ICU hospitalization (2 months maximum)
  Simple numeric rating scale for dyspnea (Dyspnea- Visual Analogic Scale (VAS)) and simple numeric rating scale assessing relief of dyspnea from 0 to 10 cm, 0 means 'no relief, no impression of improvement in breathlessness' and 10 means 'extraordinarily relieved,' performed 60 minutes after extubation and at 24 hours, dyspnea if Dyspnea-VAS > 4

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Médecine Intensive-Réanimation Hôpital Tenon, AP-HP, Paris, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided